CLINICAL TRIAL: NCT00191763
Title: Phase II Trial of Gemcitabine and Cisplatin as Neo-Adjuvant Chemotherapy for Operable Non-Small Cell Lung Cancer
Brief Title: Neo-Adjuvant Gemcitabine and Cisplatin in Treating Patients With Early Stage of Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7138; B9E-VI-S314
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2007-11-06 (Estimated); Status verified 2007-11

CONDITIONS: Carcinoma, Non-Small-Cell-Lung Cancer
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung | interventions — Gemcitabine; Cisplatin

INTERVENTIONS:
Drug: Gemcitabine
Drug: cisplatin

SUMMARY:
Based on available data, the concept of neo-adjuvant chemotherapy seems to be promising for patients with resectable non-small cell lung cancer. The exploration of new drugs and regimens are warranted. Therefore the aim of this study is to evaluate the clinical response rate of neo-adjuvant chemotherapy with gemcitabine and cisplatin in patients with operable non-small cell lung cancer stage IB, IIA-B, IIIA.

ELIGIBILITY:
Inclusion Criteria:

* define histologic or cytologic diagnosis of non small cell lung cancer.
* determine the presence of clinical Stage IB, IIA-B or IIIA disease in accordance with the revision by Mountain CF of American Joint Committee on Cancer.
* define performance status of 0-1 on ECOG scale
* do not have any prior tumor therapy
* to be suitable for curative resection

Exclusion Criteria:

* to have any treatment within the last 30 days with any investigational drug.
* to get concurrent administration of any other tumor therapy
* to be pregnant
* to have poorly controlled diabetes mellitus
* to have serious concomitant disorders.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52
Dates: Start 2002-11; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the clinical response rate of neo-adjuvant chemotherapy with gemcitabine and cisplatin in patients with operable non small cell lung cancer

SECONDARY OUTCOMES:
To evaluate the safety of neo-adjuvant chemotherapy with gemcitabine / cisplatin
To determine the complete tumor resection rate
To evaluate overall survival and time to documented disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon-Fri from 9AM to 5PM Eastern time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Istanbul, Turkey (Türkiye)

REFERENCES:
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com